CLINICAL TRIAL: NCT00965926
Title: A Pharmacokinetic Study in Healthy Non-elderly Male and Female Volunteers to Investigate the Effect of Food on the Pharmacokinetics of YM178
Brief Title: A Study to Investigate the Food Effect on the Pharmacokinetics of YM178 in Healthy, Non-elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 178-CL-078
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Volunteer; Pharmacokinetics of YM178
Keywords: Overactive Bladder; Urinary incontinence; YM178; mirabegron
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose group (Experimental): 3 way cross-over. Fasting, normal diet and high-fat diet
  Interventions: Drug: YM178
- High dose group (Experimental): 3 way cross-over. Fasting, normal diet and high-fat diet
  Interventions: Drug: YM178

INTERVENTIONS:
Drug: YM178 — oral
  Other Names: mirabegron

SUMMARY:
The purpose of the study is to evaluate the effect of food intake on the pharmacokinetics of YM178 in healthy, non-elderly adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as judged by the investigator/subinvestigator based on the results of physical examinations and all lab tests
* Body weight (at screening); female ≥40.0 kg, <70.0 kg, male ≥50.0 kg, <80.0 kg
* BMI (at screening): ≥17.6, <26.4
* Written informed consent has been obtained

Exclusion Criteria:

* Received any investigational drugs within 120 days before the screening test
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days before the screening test
* Received medication within 7 days before hospital admission or is scheduled to receive medication
* Females who are lactating, pregnant, potentially child-bearing, or willing to get pregnant during the study period
* History of drug allergies
* Upper gastrointestinal disease (e.g. nausea, vomiting, stomachache) within 7 days before hospital admission

Ages: 20 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of unchanged YM178 | Up to 96 hours post dose

SECONDARY OUTCOMES:
Urinary concentration of unchanged YM178 | Up to 96 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kantou, Japan